CLINICAL TRIAL: NCT04053829
Title: A Phase 2 Study to Investigate the Feasibility and Acceptability of the HOLOBalance System Compared to Standard Care in Older Adults at Risk for Falls: a Multi-site Study
Brief Title: Feasibility and Acceptability of HOLOBalance Compared to Standard Care in Older Adults at Risk for Falls
Acronym: HOLOBALANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University College, London (Other); Horizon 2020 - European Commission (Other); University of Ioannina (Other); Roessingh Research and Development (Other); University of Athens (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 76957
Record Dates: First submitted 2019-07-26; First posted 2019-08-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Accidental Falls; Aging; Vestibular Disorder
Keywords: Rehabilitation; Tele-rehabilitation; Physical Therapy; Coaching; Physical Activity
MeSH Terms: conditions — Vestibular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: This multi-centre, assessor-blinded, randomised proof of concept study will explore the acceptability and feasibility of providing a home-based balance tele-rehabilitation programme to older adults at risk for falls. It will 1) compare acceptability of the tele-health programme (e.g. compliance, drop-out rate) to an established home exercise programme (the OTAGO HEP) and 2) explore trends for effectiveness across a number of validated outcome measures to explore whether a future trial is warranted, and if so to provide data for a sample size estimate.
  Data will be collected at baseline (week 0) and at completion of the intervention (week 9). The flow of participants through the trial will be recorded in compliance with the CONSORT statement. The blinded outcome assessor will collect all measures at baseline and follow up and will be asked to record any incidences of unblinding and detail how this occurred.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor will be masked in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOLOBalance (Experimental): The experimental arm will use the HOLOBalance tele-rehabilitation system to provide the intervention. Participants will be required to use the HOLOBalance system on a daily basis for the duration of the 8 week study. Although participants will have daily interaction with the HOLOBalance system, they will be free to choose when to complete their exercises.
  Interventions: Device: HOLOBalance
- OTAGO Home Exercise Programme (Active Comparator): The comparator for this study is the OTAGO home exercise programme. The OTAGO is a systematic, progressive strength and balance training programme and is supported by a comprehensive workbook that provides written and pictorial instructions for each exercise. The OTAGO is well-established and is widely used in clinical practice in the UK for the management of older adults who fall or have increased risk for falling. It has been shown to be well tolerated in older adults in community settings with good adherence rates, and reduces falls rate in older adults by 35%, with greatest effects observed in frailer older women
  Interventions: Other: OTAGO Home Exercise Programme

INTERVENTIONS:
Device: HOLOBalance — The HOLOBalance tele-rehabilitation system will be used to deliver an evidence based, multi-sensory balance rehabilitation programme to participants, and will deliver a series of exercises prescribed by an expert balance physiotherapist following an initial balance assessment.
  The HOLOBalance system will use a head mounted augmented reality display to deliver exercises and games to participants and will record task performance via a combination of body worn sensors and a depth camera. The HOLOBalance tele-rehabilitation system will provide feedback to the supervising clinical team regarding task performance, participant usage and user feedback. The system will have daily presence in the users' home with users expected to complete their prescribed rehabilitation on a daily basis, which mirrors the prescribed exercise routines often provided by balance physiotherapists.
  Arms: HOLOBalance
Other: OTAGO Home Exercise Programme — The OTAGO is a systematic, progressive strength and balance training programme and is supported by a comprehensive workbook that provides written and pictorial instructions for each exercise. It is well-established and widely used in clinical practice in the UK, and has been shown to reduce falls rate in older adults by 35-40%. It is well tolerated in older adults in community settings with good adherence rates.The OTAGO has also been used as the standard intervention in previous investigations of MSR interventions in older adults. To match intervention and control interventions, participants in the OTAGO group will be asked to complete the OTAGO programme every day for the duration of the 8 week programme.
  Arms: OTAGO Home Exercise Programme

SUMMARY:
This study will utilise an assessor blinded, randomised controlled design to investigate the acceptability and feasibility of providing a novel tele-rehabilitation balance training system (HOLOBalance) for community dwelling older adults at risk for falls. Older adults (age 65-80) who meet the inclusion criteria (e.g. independently living, no neurological conditions) will be recruited from falls services and from the wider community (via AgeUK) and will be randomly allocated to receive either a prescribed exercise programme delivered by: 1) the HOLOBalance tele-rehabilitation system or 2) an exercise booklet (The OTAGO Home Exercise Programme). Participants will be required to perform a series of prescribed exercises each day (duration of up to 30 minutes per day) for the entirety of the 8-week exercise programme. These exercises will be provided via the HOLOBalance tele-rehabilitation system (intervention arm) or by written instructions (control arm).

Primary objectives for this study are to assess recruitment rate, compliance with exercise programmes (exercise diaries) and drop-out rates within the intervention group and a control group undertaking standard practice, home based balance rehabilitation (the OTAGO Home Exercise Programme) to explore whether HOLOBalance is acceptable to participants. Furthermore, acceptability to older adults will also be investigated via exit interviews performed within the HOLOBalance tele-rehabilitation intervention arm.

Feasibility will be assessed by documenting adverse events (and SAE's), adverse device effects (and SADE's), deviations from protocol and feedback from treating clinicians. Implementation issues such as technology break down, service delivery and usability issues will also be documented. Secondary outcomes to explore trends for effectiveness will investigate performance of both groups at baseline and after the 8 week intervention across a range of outcome measures associated with balance function and falls risk, cognitive function, Physical activity and social participation, and subjective report of mobility and balance.

ELIGIBILITY:
Inclusion Criteria:

* Independent community-dwelling participants able to walk 500 meters independently or with a stick
* No significant visual impairment
* Able to understand and to consent to the research
* A score of >22 on the MoCA, i.e. adults with no or mild cognitive impairment;
* At risk of falls (i.e. FGA less than 22/30), have significant fear of falling (FESI short form >10) or having experienced a fall/s in the last 12 months
* Willing to participate and to comply with the proposed training and testing regime.
* Available space of 1x2 metres at home and sufficient home broadband to allow the system to operate as designed

Exclusion Criteria:

* Orthostatic hypotension or uncontrolled hypertension
* Have depression i.e. a score of >10 at the Geriatric depression scale
* Have cognitive impairment as indicated by the MoCA score(score <22)
* Other neurological problem (stroke, Parkinson's, peripheral neuropathy)
* Acute musculo-skeletal injury that prevents participation in a structured exercise programme (e.g. lower limb fracture)
* No internet connection at home
* Has participated in a clinical drug trial in the past 6 months
* Currently receiving falls and/or cognitive rehabilitation.
* Has an implanted medical device or cardiac pacemaker

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Acceptability Assessment 1: Recruitment Rate | Through study completion (12 months)
  Assessment of recruitment rate of study (% of eligible participants enrolled)
Acceptability Assessment 2: Programme Compliance | Through study completion (12 months)
  Comparison of compliance with exercise programmes (% of sessions completed) within the intervention group and a control group undertaking standard practice, home based balance rehabilitation (the OTAGO Home Exercise Programme).
Acceptability Assessment 3: Drop out rate | Through study completion (12 months)
  Comparison of drop-out rates (%) between the intervention group and a control group undertaking standard practice, home based balance rehabilitation (the OTAGO Home Exercise Programme).
Acceptability 4: Qualitative interview | Collected at end of each participants participation in the study (After 8 weeks)
  Acceptability of HOLOBalance to older adults will be investigated via exit interviews performed within the tele-rehabilitation intervention arm.
Feasibility of providing HOLOBalance 1: Monitoring of Adverse and Serious Adverse Events | Through study completion (12 months)
  Feasibility will be assessed by documenting adverse events (and SAE's) and adverse device effects (and SADE's).
Feasibility of providing HOLOBalance 2: Monitoring for deviations from study protocol | Through study completion (12 months)
  Assessment of any deviations from protocol reported logged in the site files using the deviation from protocol form.

SECONDARY OUTCOMES:
Balance Function Assessment | Baseline (Week 0) and Follow up (Week 9)
  Functional Gait Assessment. This is a 10-item test that assesses performance on complex gait tasks (e.g. walking with head turns or stopping and turning). Each item is rated on a 4 point scale (0-3) with higher scores indicating better task performance.
Balance Function Assessment | Baseline (Week 0) and Follow up (Week 9)
  Mini-BESTest. This is a 14-item test that assesses dynamic balance components including anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. The 14 items are scored on a 3 point scale (0-2), with a maximum score of 28 points awarded. Higher scores indicate better task performance.
Cognitive Function Assessment | Baseline (Week 0) and Follow up (Week 9)
  Montreal Cognitive Assessment. This test includes sections on visuospatial/executive function (alternating trail-making, cube copy, clock drawing), naming (lion, rhinoceros, camel), attention (forward and backward digit span, tapping to the letter A, subtracting 7s from 100), language (sentence repetition, letter fluency), abstraction (similarities between train and bicycle, watch and ruler), memory (delayed verbal recall of 5 words) and orientation to time and place (6 questions)
Cognitive Function Assessment | Baseline (Week 0) and Follow up (Week 9)
  Cambridge Neuropsychological Test Automated Battery (CANTAB). The test battery includes: (i) Motor screening task to assess a participant's general ability to understand and complete tasks and highlights if any sensorimotor or hearing impairments will have an impact on test performance, (ii) Paired Associated Learning assesses visual associative learning and memory, (iii) Spatial Working Memory to assess one's ability to retain and use visuospatial input, (iv) Reaction Time tests a person's mental and motor response speed, (v) Rapid Visual Information Processing assesses the ability to maintain visual attention and continuous performance on a task and (vi) Delayed Matching to Sample tests visual recognition memory and short term visual memory.
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  Rapid Assessment of Physical Activity (RAPA). This is a 9-item, self-administered questionnaire developed to provide an easily administered and interpreted means of assessing levels of physical activity among adults older than 50 years. RAPA evaluates a wide range of physical activity level, from sedentary to vigorous activity, as well as strength and flexibility training
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  WHO Disability Assessment Schedule 2.0. This is an assessment which provides a global measure of disability. It covers the following domains of functioning: Cognition - understanding & communicating; Mobility- moving & getting around; Self-care- hygiene, dressing, eating & staying alone; Getting along- interacting with other people; Life activities- domestic responsibilities, leisure, work & school; Participation- joining in community activities.
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  Activities-Specific Balance Confidence Scale (ABC). This questionnaire assesses patients perceived confidence for performing 16-activities of daily living without losing balance. Scores ≤67/100% indicate increased falls risk.
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  Falls Self-Efficacy Scale International. This is a short, easy to administer tool measuring an individual's level of concern regarding falling during social and physical activities inside and outside the home, whether or not the person actually does the activity. Level of concern is measured on a four-point Likert scale (1=not at all to 4=very). It has excellent internal validity and test-retest reliability. Scores of >23 for the long form and >10 for the short form have been suggested as cut points for indicating high concern about falling
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  Behavioral Regulation in Exercise Questionnaire (BREQ-3). This is a 24 item questionnaire to assess motivation to exercise. Participants rate whether statements apply to themselves (or not) using a 5 point likertLikert scale ranging from 0 (Not true for me) to 4 (Very true for me)
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  EQ-5D-5L. This is a standardized, valid and reliable simple, generic measure of health status for clinical and economic appraisal. The EQ-5D-5L has 5 dimensions (mobility, selfcare, usual activities, pain/discomfort, anxiety/depression) and includes the EQ visual Analogue scale (EQ VAS). The respondent is asked to rate their health status on these five dimensions from 1 to 5 respectively as no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeledlabelled 'the best health you can imagine' and 'the worst health you can imagine'. The respondent is asked to mark an X on the scale to indicate "how your health is TODAY".
Subjective Questionnaire | Baseline (Week 0) and Follow up (Week 9)
  Environmental Mobility Scale. This is a self-report scale assessing the effect of the physical environment on community mobility. Twenty-four features of the physical environment are identified. For each feature, an encounter question (How often do you?) is paired with an avoidance question (How often do you avoid?). Subjects report on frequency of encounter and avoidance behaviour using a five-point ordinal scale (never, rarely, sometimes, often, always). The test-retest reliability of the questionnaire is good.

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, PhD, Principal Investigator — University College, London; Marousa Pavlou, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Electronic data will be anonymised and uploaded to a data repository that supports restricted access.Restricted access will be required for the data generated from the study participants.These files will not be made publicly available and sharing will be made possible only by the approval of the Holobalance data management board, and use and re-use of the pilot dataset will be subject to the license under which the data objects were deposited.
  Holobalance will also consider to deposit the content under an embargo status and provide an end date for the embargo in order to explore exploitation possibilities which affect the availability of data for third parties and usually is not finalized before the end of the project and the outcomes of the pilot study.
Supporting Information: Study Protocol
Time Frame: Upon completion of all project outcomes and assessments for commercial exploitation.
Access Criteria: Sharing will be made possible only by the approval of the Holobalance data management board, and use and re-use of the pilot dataset will be subject to the license under which the data objects were deposited.

REFERENCES:
- [Derived] Tsakanikas V, Gatsios D, Pardalis A, Tsiouris KM, Georga E, Bamiou DE, Pavlou M, Nikitas C, Kikidis D, Walz I, Maurer C, Fotiadis D. Automated Assessment of Balance Rehabilitation Exercises With a Data-Driven Scoring Model: Algorithm Development and Validation Study. JMIR Rehabil Assist Technol. 2022 Aug 31;9(3):e37229. doi: 10.2196/37229. PMID 36044258
- [Derived] Liston M, Genna G, Maurer C, Kikidis D, Gatsios D, Fotiadis D, Bamiou DE, Pavlou M. Investigating the feasibility and acceptability of the HOLOBalance system compared with standard care in older adults at risk for falls: study protocol for an assessor blinded pilot randomised controlled study. BMJ Open. 2021 Feb 12;11(2):e039254. doi: 10.1136/bmjopen-2020-039254. PMID 33579762
- See also: HOLOBalance study website — http://holobalance.eu